CLINICAL TRIAL: NCT03275987
Title: A Population-based Randomized Trial to Promote Cancer Screening Among Unscreened Medicaid Recipients in Minnesota
Brief Title: Promoting Cancer Screening Among Medicaid Recipients in Minnesota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minnesota Department of Health (Other Government)
Responsible Party: Principal Investigator, Jonathan Slater, Chief of Cancer Control Section, Minnesota Department of Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Innovations2017
Record Dates: First submitted 2017-09-01; First posted 2017-09-08 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Colorectal Cancer; Breast Cancer
Keywords: cancer screening
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mammography treatment (Experimental): Mammography direct mail coupled with a financial incentive
  Interventions: Behavioral: Mammography direct mail coupled with a financial incentive
- Mammography control/delayed intervention (Active Comparator): Usual care (for 15 months); Mammography direct mail coupled with financial incentive (after 15 months)
  Interventions: Behavioral: Mammography direct mail coupled with a financial incentive; Behavioral: Usual care
- Colonoscopy treatment (Experimental): Colonoscopy direct mail coupled with a financial incentive
  Interventions: Behavioral: Colonoscopy direct mail coupled with a financial incentive
- Colonoscopy control/delayed intervention (Active Comparator): Usual care (for 15 months); Colonoscopy direct mail coupled with financial incentive (after 15 months)
  Interventions: Behavioral: Usual care; Behavioral: Colonoscopy direct mail coupled with a financial incentive

INTERVENTIONS:
Behavioral: Mammography direct mail coupled with a financial incentive — The intervention groups received innovative and persuasive direct mail materials coupled with an incentive for using their Medicaid benefit to get screened.
  Arms: Mammography control/delayed intervention; Mammography treatment
Behavioral: Usual care — Group received usual care, and direct mail 15 months after treatment group received intervention.
  Arms: Colonoscopy control/delayed intervention; Mammography control/delayed intervention
Behavioral: Colonoscopy direct mail coupled with a financial incentive — The intervention groups received innovative and persuasive direct mail materials coupled with an incentive for using their Medicaid benefit to get screened.
  Arms: Colonoscopy control/delayed intervention; Colonoscopy treatment

SUMMARY:
This study evaluates the effectiveness of persuasive direct mail materials coupled with an incentive for increasing breast and colorectal cancer screening among people enrolled in Medicaid. Half of age- and gender-appropriate enrollees received this intervention; the other half received the same intervention 15 months later

DETAILED DESCRIPTION:
This trial was conducted between April 2014 and July 2015 and implemented through Sage, the National Breast and Cervical Cancer Early Detection Program (NBCCEDP) in Minnesota and housed within the Minnesota Department of Health (MDH). The target population was all Minnesota Medicaid recipients ages 50-74 overdue for breast cancer and colorectal cancer screening. Claims data, obtained from MDHS, were used to determine patient characteristics and outcomes. Individuals who were not enrolled in Medicaid, who were not overdue for BC or CRC screening, or who were not in the 50-74 age range were excluded prior to analysis.

To determine the efficacy of the interventions we used a two group posttest-only randomized design with all eligible MA beneficiaries randomly assigned to one of two groups: Direct Mail plus Incentive (with patient navigation) versus usual care.

The primary outcomes were completion of mammography or colonoscopy within 12 weeks after implementation of the intervention. Current Procedural Technology (CPT) codes from Medicaid claims data were used to determine if an individual had received either mammography or colonoscopy. Specific CPT codes used for mammography were conventional mammography (77055-77057), digital mammography (G0202, G0204, G0206), and computer-aided detection mammography (77051, 77052). CPT codes used for colonoscopy were G0105, G0121, 45378, and 45380-45385. Mammography and colonoscopy outcomes were measured dichotomously. Outcomes were based on the presence of screening mammography and colonoscopy claims occurring for 10 weeks after the first mailings.

The mammography and colonoscopy interventions were examined separately. Across treatment and control, study sample characteristics were compared and absolute differences were assessed using t-test and χ2 statistics. Main outcome analyses consisted of logistic regression to compute odds ratios for receiving mammography or colonoscopy and for covariate adjustment. Two separate logistic regression models were examined for both mammography and colonoscopy interventions: (1) a bivariate model that examined treatment versus control, and 2) a multivariate model that adjusted for covariates. All analyses were conducted using Stata, version 13.

Some individuals lost Medicaid coverage on a monthly basis during the study period, and others had inaccurate mailing addresses (< 2% of each study sample). Therefore not everyone received the treatment as intended, and individuals that received the intervention may not have had Medicaid claims available post-intervention. Our outcome analyses were intent-to-treat analyses that included all individuals randomized to treatment or control groups at initiation of intervention regardless of whether they lost coverage post-randomization or if they had an inaccurate mailing address.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in Minnesota Medicaid for at least the prior year

Exclusion Criteria:

* Younger than 50 or older than 74
* Women having mammogram in 15 months before trial (mammography intervention)
* Evidence of a colonoscopy in the past 10 years, flexible sigmoidoscopy in the past five years, or fecal immunochemical or fecal occult blood test in the past year (colonoscopy intervention)

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Mammography arm was limited to women. Colonoscopy arm included both genders.
Enrollment: 138554 (Actual)
Dates: Start 2014-04-23 (Actual); Primary Completion 2014-09-30 (Actual); Study Completion 2017-05-10 (Actual)

PRIMARY OUTCOMES:
screening mammography or colonoscopy | Within 12 weeks of first mailing
  Evidence of a mammogram received after implementation of the intervention, based on presence of CPT codes in Medicaid claims data set.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S Slater, PhD, Principal Investigator — Minnesota Department of Health; Christina L Nelson, MS, Study Director — Minnesota Department of Health
Locations (1):
- Minnesota Department of Health, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No